CLINICAL TRIAL: NCT05894486
Title: Phase II Study to Evaluate the Efficacy and Safety of 177Lu-Dotatate in the First-line Treatment of Inoperable Patients With Locally Advanced or Metastatic, Somatostatin Receptor-positive G2 or G3 Gastroenteropancreatic Neuroendocrine Tumors
Brief Title: Phase II Study to Evaluate the Efficacy and Safety of 177Lu-Dotatate in the First-line Treatment of Patients With Locally Advanced or Metastatic, Somatostatin Receptor-positive G2 or G3 Gastroenteropancreatic Neuroendocrine Tumors
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XT-XTR008-2-01
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Neuroendocrine Tumors
Keywords: PRRT; Lutetium[177Lu]
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — lutetium Lu 177 dotatate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lutetium[177Lu] Oxodotreotide Injection (Experimental): Treatment consisted of a cumulative administered radioactivity of 29.6 Giga Becquerel (GBq) (800 mCi) Lutetium[177Lu] Oxodotreotide Injection: Four administrations of 7.4 GBq (200 mCi).
  Concomitant amino acids were given with each administration for kidney protection.
  Lutetium[177Lu] Oxodotreotide Injection was administered at 8 +/- 1-week intervals, which could be extended up to 16 weeks to accommodate resolving acute toxicity.
  In case participants experienced clinical symptoms (i.e. diarrhoea and flushing) associated with their carcinoid tumours, Octreotide s.c. rescue injections were allowed.
  Interventions: Drug: Lutetium[177Lu] Oxodotreotide Injection

INTERVENTIONS:
Drug: Lutetium[177Lu] Oxodotreotide Injection — Lutetium[177Lu] Oxodotreotide InjectionFour administrations of 7.4 GBq (200 mCi) Lutetium[177Lu] Oxodotreotide Injection administered at 8 +/- 1-week intervals, which could be extended up to 16 weeks to accommodate resolving acute toxicity
  Other Names: 177Lu-DOTA0-Tyr3-Octreotate

SUMMARY:
his was a single-center, single-arm phase II study evaluate the efficacy and safety of Lutetium[177Lu] Oxodotreotide Injection in the first-line treatment of unresectable or metastatic, progressive, G2 or G3, somatostatin receptor positive gastroenteropancreatic neuroendocrine tumours.

DETAILED DESCRIPTION:
After the screening period, participants who signed the ICF and were eligible for the study in accordance with the entry criteria were assigned to treatment with Lutetium[177Lu] Oxodotreotide Injection. Objective tumor assessment in both groups was performed every 12+/-1 weeks from the first treatment date according to RECIST 1.1 Criteria until progression.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and willingness to sign a written informed consent document.
2. Aged 18-75 years.
3. Histopathologically confirmed G2 or G3 unresectable locally advanced or metastatic GEP-NET, Ki67 index ≥10 and ≤ 55%. (based on the fifth edition of the WHO classification and grading criteria for neuroendocrine， tumors of the digestive system in 2019, to be centrally confirmed).
4. Subjects have not received prior systemic antitumor therapy for the current stage of NET.
5. Presence of at least 1 measurable site of disease (based on RECIST 1.1).
6. All target lesions (based on RECIST 1.1) at baseline must be confirmed as growth inhibitor receptor positive by 68Ga-Dotatate PET/CT.
7. ECOG score of 0 or 1.
8. Subjects of childbearing potential voluntarily use an effective method of contraception, such as condoms, oral or injectable contraceptives, IUDs, etc., during treatment and within 3 months of the last use of the trial drug.

Exclusion Criteria:

1. Serum creatinine >150 μmol/L (1.7 mg/dL) or creatinine clearance <50 ml/min (Cockcroft Gault formula).
2. Hemoglobin <80g/L, or white blood cell count <2.0×109/L, or platelets <75×109/L.
3. Serum total bilirubin > 3 × upper limit of normal (ULN).
4. Serum albumin <30g/L.
5. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5×ULN.
6. International normalized ratio (INR) > 1.5 or partially activated prothrombin time (APTT) > 1.5 x ULN.
7. Pregnant or lactating females.
8. Received peptide receptor radionuclide therapy(PRRT) prior to randomization.
9. Received the following treatments within 4 weeks prior to treatment, including but not limited to surgery (except biopsy), radical radiotherapy, hepatic artery interventional embolization, cryoablation of liver metastases, or radiofrequency ablation.
10. Received systemic antitumor therapy such as targeted therapy, immunotherapy, antitumor herbal therapy, chemotherapy within 4 weeks prior to randomization.
11. Toxicity of prior antitumor therapy has not returned to ≤ grade 1 levels (except for alopecia).
12. Received external beam radiation therapy for bone metastases within 2 weeks prior to treatment.
13. More than 25% of bone marrow with prior external radiation radiotherapy.
14. Known brain metastases, unless these metastases have been treated and stabilized for at least 24 weeks, prior to enrollment in the study.
15. Uncontrolled congestive heart failure.
16. uncontrolled diabetes mellitus, including baseline fasting glucose > 2 x ULN.
17. Any patient receiving treatment with short-acting Octreotide, which cannot be interrupted for 24 h before and 24 h after the administration of Lutetium[177Lu] Oxodotreotide Injection, or any patient receiving treatment with Octreotide LAR, which cannot be interrupted for at least 6 weeks before the administration of Lutetium[177Lu] Oxodotreotide Injection.
18. Known other malignancies (except for those without recurrence within 5 years after adequate treatment)
19. Known hypersensitivity to Lutetium[177Lu] Oxodotreotide Injection or oxytetracycline acetate microsphere components and their excipients.
20. Known to be unsuitable for enhanced CT or MRI contrast imaging due to allergic reaction or renal insufficiency
21. Any clinically significant active infection, including Positive human immunodeficiency virus (HIV) antibody.
22. Positive for hepatitis B virus (HBV) surface antigen (HBsAg) and positive for HBV DNA (≥1×104 copies/ml or judged positive by research center criteria), or positive for hepatitis C virus (HCV) antibodies.
23. Participated in other drug clinical trials within 4 weeks prior to the first treatment and received treatment with the corresponding trial drug.
24. Any other disease, mental status or surgical condition that is uncontrolled, may interfere with study completion (including poor compliance) or is inappropriate for the use of the investigational drug.
25. Other treatment options (e.g., chemotherapy, targeted therapy) that, in the opinion of the investigator, are more appropriate for the patient than the treatment provided in the study based on the patient's disease characteristics, i.e., the investigational drug is not the best therapeutic agent for clinical practice.
26. Subjects who, in the judgment of the investigator, are suspected of having a disease or condition that makes them unsuitable for the study drug disease or condition.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-05 (Estimated); Primary Completion 2025-06-05 (Estimated); Study Completion 2026-06-05 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 in all participants | Up to 2 years
  ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1. For this analysis, ORR will be assessed in all participants

SECONDARY OUTCOMES:
Incidence of Treatment-Related Adverse Events | Until 30 days after the last treatment
  An AE was defined as any untoward medical occurrence in a participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment. The number of participants who experienced ≥1 AE will be presented.
Progression-free Survival (PFS) per RECIST 1.1 in all participants | Up to 2 years
  PFS is defined as the time from the date of first dose to the first documented disease
Disease control rate(DCR) | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China